CLINICAL TRIAL: NCT04481698
Title: Mesoglycan for Pain Control After Open Excisional HAEMOrrhoidectomy (MeHAEMO): An Observational Multicentre Study on Behalf of the Italian Society of Colorectal Surgery (SICCR)
Brief Title: Mesoglycan for Pain Control After Open Excisional HAEMOrrhoidectomy
Acronym: MeHAEMO
Status: Completed | Type: Observational
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Collaborators: Gaetano Gallo (Unknown); Giuseppe Sammarco (Unknown); Giuseppe Clerico (Unknown); Alessandro Sturiale (Unknown); Michele Manigrasso (Unknown); Alberto Realis Luc (Unknown); Mario Trompetto (Unknown)
Responsible Party: Sponsor
Other Study IDs: 176/2017
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Haemorrhoidal Disease; Post-operative Pain; Thrombosis
MeSH Terms: conditions — Pain, Postoperative; Thrombosis | interventions — mesoglycan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mesoglycan: All patients received the standard post-operative therapy (a recommended oral dose of ketorolac tromethamine of 10 mg every 4-6 hours, not exceeding 40 mg per day and not exceeding 5 post-operative days according to the indications for short-term management of moderate/severe acute post-operative pain and stool softeners) plus mesoglycan (Prisma® 30 mg 2 vials i.m./day for the first 5 post-operative days and then Prisma® 50 mg 1 oral tablet twice/day for an additional 30 days, Mediolanum Farmaceutici, Milan, Italy)
  Interventions: Other: Mesoglycan
- Control: standard post-operative therapy (a recommended oral dose of ketorolac tromethamine of 10 mg every 4-6 hours, not exceeding 40 mg per day and not exceeding 5 post-operative days according to the indications for short-term management of moderate/severe acute post-operative pain and stool softeners)
  Interventions: Other: Mesoglycan

INTERVENTIONS:
Other: Mesoglycan — Prisma® 30 mg 2 vials i.m./day for the first 5 post-operative days and then Prisma® 50 mg 1 oral tablet twice/day for an additional 30 days

SUMMARY:
Haemorrhoidal disease (HD) is the most common proctological disease, with a prevalence that can reach up to 39% of the population. Although I and II degree HD can be treated successfully with medical therapy or office-based procedures , excisional haemorrhoidectomy remains the gold standard technique in patients with III and IV degree HD, obtaining a much lower rate of recurrence than non-excisional methods, such as Doppler-guided haemorrhoidal artery ligation or stapled haemorrhoidopexy. However, both open and closed haemorrhoidectomies are associated with a significant rate of post-operative pain , which may be due to the incorporation of sensitive anal mucosa and fibres of the internal sphincters during the ligation of the vascular pedicle, post-operative scars, hygiene/social habits, hard stool, or oedema of the necessary mucocutaneous bridge.

Regarding the oedema/thrombosis of the mucocutaneous bridges, we strongly believe that it is the main cause of post-operative pain, and we have shown that the use of mesoglycan, a polysaccharide complex with antithrombotic and profibrinolytic properties, can reduce the rate of post-operative thrombosis and consequently post-operative pain 7-10 days after the procedures, improving patient quality of life and speeding up the recovery of daily activities.

Furthermore, its usefulness is also evident in the treatment of the acute phase of external haemorrhoidal thrombosis.

The aim of the study was to evaluate the efficacy of mesoglycan in the post-operative period of patients who underwent open excisional diathermy haemorrhoidectomy, confirming the previously obtained results

DETAILED DESCRIPTION:
This was a retrospective multicentre study and is reported according to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement for cohort studies

Between September and December 2017, 206 patients with III and IV degree HD, according to Goligher classification, from sixteen colorectal referral centres belonging to SICCR (Società Italiana di Chirurgia Colorettale), who satisfied inclusion criteria underwent open excision haemorrhoidectomy.

The results obtained were compared with a homogeneous sample of 192 patients who underwent OEH in the same centres between April and July 2017 and who had received standard post-operative therapy without mesoglycan.

All patients received the standard post-operative therapy (a recommended oral dose of ketorolac tromethamine of 10 mg every 4-6 hours, not exceeding 40 mg per day and not exceeding 5 post-operative days according to the indications for short-term management of moderate/severe acute post-operative pain and stool softeners) plus mesoglycan (Prisma® 30 mg 2 vials i.m./day for the first 5 post-operative days and then Prisma® 50 mg 1 oral tablet twice/day for an additional 30 days, Mediolanum Farmaceutici, Milan, Italy).

In each referral centre, the procedures were carried out by an experienced surgeon who had performed more than 200 haemorrhoidectomies.

A clinical external examination was performed the first post-operative day, and an anorectal digital evaluation with proctoscopy was performed at T2, T3 and T4.

During each follow-up visit, post-operative pain was evaluated at rest, after defecation and after anorectal digital examination using a visual analogue scale (minimum score = 0; maximum score = 10).

Quality of life was evaluated pre- and post-operatively 90 days after the procedure using the SF-12 questionnaire.

Polypharmacy was defined as 5 or more medications daily. Thrombosis was defined as one or more swollen painful piles at the site of the mucocutaneous bridge and was assessed at T2, T3 and T4.

Surgical wound healing (granulation) was evaluated at T2, T3 and T4 using the following 3 items: infected, granulating, healed.

Autonomy was evaluated at T2, T3 and T4 using the following 4 items: complete inactivity, total autonomy at home, ability to drive, return to normal activities (autonomy at home, driving, working).

Bowel movements were evaluated, according to the proper guidelines, at T2, T3 and T4, and patients were classified in three categories: regular, constipation or diarrhoea.

ELIGIBILITY:
Inclusion Criteria:

* III and IV degree Hemorrhoidal Disease
* Age > 18
* Written Informed Consent

Exclusion Criteria:

* Age <18
* Past or present history of:
* Coagulopathy
* Cardiac Diseases
* Anticoagulant Therapies
* Colorectal or Anal Neoplasms
* Inflammatory Bowel Disease
* Pelvic Radiotherapy
* Anal Surgery
* Allergy to Mesoglycan
* Inability to return for post-operative control visits

Age Groups: Child, Adult, Older Adult
Study Population: All patients received the standard post-operative therapy (a recommended oral dose of ketorolac tromethamine of 10 mg every 4-6 hours, not exceeding 40 mg per day and not exceeding 5 post-operative days according to the indications for short-term management of moderate/severe acute post-operative pain and stool softeners) plus mesoglycan (Prisma® 30 mg 2 vials i.m./day for the first 5 post-operative days and then Prisma® 50 mg 1 oral tablet twice/day for an additional 30 days, Mediolanum Farmaceutici, Milan, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in Post-operative Pain | Day 7, Day 20, Day 40
  VAS

SECONDARY OUTCOMES:
Changes in post-operative Thrombosis | Day 7, Day 20, Day 40
  Dichotomous parameter (Yes or Not)
Changes in post-operative Bleeding | Day 7, Day 20, Day 40
  Dichotomous parameter (Yes or Not)
Quality of Life (QoL) | pre- and post-operatively 90 days after the procedure
  We used the 12-Item Short Form Survey (SF-12) to assess QoL
Changes in Surgical Wound Healing | Day 7, Day 20, Day 40
  we evaluated wound healing with the following scale: infected, granulating, healed
Changes Autonomy | Day 7, Day 20, Day 40
  we evaluated autonomy with the following parameters: complete inactivity (patient unable to performing any activity), total autonomy at home, ability to drive, return to normal activities (patient able to performing any activity)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Gallo G, Martellucci J, Sturiale A, Clerico G, Milito G, Marino F, Cocorullo G, Giordano P, Mistrangelo M, Trompetto M. Consensus statement of the Italian society of colorectal surgery (SICCR): management and treatment of hemorrhoidal disease. Tech Coloproctol. 2020 Feb;24(2):145-164. doi: 10.1007/s10151-020-02149-1. Epub 2020 Jan 28. PMID 31993837
- [Result] Cocorullo G, Tutino R, Falco N, Licari L, Orlando G, Fontana T, Raspanti C, Salamone G, Scerrino G, Gallo G, Trompetto M, Gulotta G. The non-surgical management for hemorrhoidal disease. A systematic review. G Chir. 2017 Jan-Feb;38(1):5-14. doi: 10.11138/gchir/2017.38.1.005. PMID 28460197
- [Result] Simillis C, Thoukididou SN, Slesser AA, Rasheed S, Tan E, Tekkis PP. Systematic review and network meta-analysis comparing clinical outcomes and effectiveness of surgical treatments for haemorrhoids. Br J Surg. 2015 Dec;102(13):1603-18. doi: 10.1002/bjs.9913. Epub 2015 Sep 30. PMID 26420725
- [Result] Gallo G, Mistrangelo M, Passera R, Testa V, Pozzo M, Perinotti R, Lanati I, Lazzari I, Tonello P, Ugliono E, De Luca E, Realis Luc A, Clerico G, Trompetto M. Efficacy of Mesoglycan in Pain Control after Excisional Hemorrhoidectomy: A Pilot Comparative Prospective Multicenter Study. Gastroenterol Res Pract. 2018 Mar 19;2018:6423895. doi: 10.1155/2018/6423895. eCollection 2018. PMID 29743886
- [Result] Bessa SS. Diathermy excisional hemorrhoidectomy: a prospective randomized study comparing pedicle ligation and pedicle coagulation. Dis Colon Rectum. 2011 Nov;54(11):1405-11. doi: 10.1097/DCR.0b013e318222b5a9. PMID 21979186